CLINICAL TRIAL: NCT00611832
Title: Evaluation of a Video-Based Media Series to Promote Effective Parenting
Acronym: ParentMedia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DA021307; R01DA021307 (NIH)
Record Dates: First submitted 2008-02-06; First posted 2008-02-11 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Childhood Disruptive Behavior Problems
Keywords: behavior problems; children; prevention; television; media; parenting
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard (Active Comparator): Standard "information-only" version of the television series that includes only modeling and demonstration of the targeted parenting skills
  Interventions: Behavioral: Triple P Media Series -- Standard "Information-Only" version
- Enhanced (Experimental): Enhanced "behavior activation" version of the television series that includes all of the content of the standard "information-only" version, but is also designed to actively promote parental behavior change, through additional content elements addressing attributions, self-efficacy and expectancies, social support, and emotional reactivity.
  Interventions: Behavioral: Triple P Media Series -- Enhanced "Behavior Activation" version
- Control (No Intervention): Waitlist control

INTERVENTIONS:
Behavioral: Triple P Media Series -- Standard "Information-Only" version — 10 episodes, 12 minutes per episode, 2 episodes viewed per week for a total of 5 weeks. Demonstrates parenting practices for effectively handling a range of difficult child behaviors.
  Arms: Standard
Behavioral: Triple P Media Series -- Enhanced "Behavior Activation" version — 10 episodes, 12 minutes per episode, 2 episodes viewed per week for a total of 5 weeks. Demonstrates parenting practices for effectively handling a range of difficult child behaviors; includes specific content elements designed to promote parents' adoption of the targeted parenting skills
  Arms: Enhanced

SUMMARY:
Researchers are developing and experimentally evaluating two variants of a 10-episode, brief (12 minutes per episode), infotainment-style television series targeted at parenting practices, to determine the potential value of television for bringing evidence-based parenting practices to parents. The study compares an "information-only" version of the television series against an "enhanced" version that is designed to actively promote parents' adoption of the targeted strategies. Both versions of the series are compared against a waitlist control group. The media series is derived from the Triple P Positive Parenting Program.

DETAILED DESCRIPTION:
The mass media, and television in particular, hold significant potential as part of a population-wide strategy for bringing evidence-based parenting practices to a broad range of parents experiencing challenges raising their children. The potential of television for affecting parenting has received very little research attention, however; thus, little is known about how media messages to affect parenting practices might be optimally designed. This study will develop and experimentally evaluate two variants of a 10-episode, brief (12 minutes per episode), infotainment-style television series targeted at parenting practices, derived from the Triple P-Positive Parenting Program (Sanders, 1999). A sample of 300 families of children ages 3-6 years with somewhat elevated disruptive behavior problems will be randomized to (a) receive a standard "information-only" version of the series that includes only modeling and demonstration of target parenting skills, (b) receive an enhanced "behavior activation" version of the series designed to actively promote parental behavior change, through elements addressing attributions, self-efficacy and expectancies, social support, and emotional reactivity, or (c) a waitlist control group. Measures of parents' parenting practices, cognitions, affect, and social support, and children's disruptive behavior problems, will be obtained at baseline, post-intervention, and 6-month follow-up. The relative efficacy of the standard and enhanced versions of the Triple P Media Series in improving these outcomes will be examined, as well as moderators of these effects, such as baseline level of behavior problems and parental stress. This study will further our understanding of the potential value of television programming for improving parenting practices.

ELIGIBILITY:
Inclusion Criteria:

* parent(s) living with a child 3 to 6 years old
* child scores 1 or more standard deviations above the mean on the Eyberg Child Behavior Inventory
* English speaking
* parent at least 20 years old

Exclusion Criteria:

* currently receiving any other structured parenting intervention (home visits, parenting classes, individual parent training, family therapy)
* father-only households

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Child problem behavior: measured by the Eyberg Child Behavior Inventory (Eyberg & Ross, 1978), phone interview, and observation coding from a structured lab task procedure | baseline, immediate post, 6-month follow-up
Problematic parenting practices: measured by the Parenting Scale (Arnold et al., 1993), phone interview, and observation coding from a structured lab task procedure | baseline, immediate post, 6-month follow-up

SECONDARY OUTCOMES:
Parent knowledge: Triple P Parenting Quiz | baseline, immediate post, 6-month follow-up
Parental attributions for child misbehavior: Parent's Attributions for Child's Behavior Measure (Pidgeon & Sanders, 2004) | baseline, immediate post, 6-month follow-up
Parental self-efficacy: Problem Behavior and Setting Checklist (Sanders & Wooley, 2005) | baseline, immediate post, 6-month follow-up
Parental stress: Depression Anxiety Stress Scale, Short Form (Lovibond & Lovibond, 1995) | baseline, immediate post, 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Carol W Metzler, PhD, Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States